CLINICAL TRIAL: NCT07338721
Title: Does Using Ultrasound Guidance During Axillary Incision Improve Sentinel Lymph Node Detection Compared to Standard Methods in Breast Cancer Patients?
Brief Title: Does Ultrasound Guidance Axillary Incision Improve Sentinel Lymph Node Detection in Breast Cancer?
Status: Recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Baris Karakas, Assoc. Prof., Antalya Training and Research Hospital
Other Study IDs: AEAH-GS-BRK-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Sentinel Lymph Node Biopsy
Keywords: Breast cancer; Axilla; Sentinel Lymph Node Biopsy; Ultrasonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The ultrasound-guided axillary incision group.: In the ultrasound-guided axillary incision group, the incision is made parallel to the Langer lines under ultrasound guidance, targeting the projection of the first lymph node at the axillary entry.
  Interventions: Procedure: Ultrasound-guided axillary incision group
- The standard hairline axillary incision group: In the ultrasound-guided axillary incision group, the incision is made at the ultrasound-identified projection of the first lymph node at the axillary entry.
  Interventions: Procedure: The standard axillary incision

INTERVENTIONS:
Procedure: Ultrasound-guided axillary incision group — In the ultrasound-guided axillary incision group, the incision is made at the ultrasound-identified projection of the first lymph node at the axillary entry.
  Groups: The ultrasound-guided axillary incision group.
Procedure: The standard axillary incision — In the standard group, the SLNB incision is made parallel to the Langer lines below the axillary hairline.
  Groups: The standard hairline axillary incision group

SUMMARY:
This single-center randomized controlled trial evaluates whether detecting the first lymph node at the axillary entrance with ultrasound guidance, followed by a targeted axillary incision over the pencil-marked projection, improves sentinel lymph node identification compared to the conventional axillary hairline landmark. The study hypothesizes that this technique enables a smaller incision, minimizes tissue dissection, and reduces operative time.

DETAILED DESCRIPTION:
Axillary lymph node status is a key prognostic factor in breast cancer treatment planning. Accurate axillary staging is essential for optimal management. Sentinel lymph node biopsy (SLNB) provides reliable nodal assessment and is associated with lower morbidity relative to axillary dissection. The sentinel lymph node is the initial recipient of lymphatic drainage from the primary tumor, and breast lymphatics typically drain into at least one sentinel node.

The majority of sentinel nodes are located in level I, particularly within the anterior axillary (pectoral) lymph nodes. These nodes are positioned at the inferolateral border of the pectoralis minor muscle, adjacent to the lateral thoracic vessels, and are typically in contact with the axillary tail of the breast.

The standard axillary incision for SLNB is performed parallel to the Langer line, below the axillary hairline. Blue-stained lymph nodes are identified and excised by following the blue-stained lymphatic channels.

The anterior axillary (pectoral) lymph node can be identified by placing the ultrasound transducer on the flattened lateral breast and axillary tail after appropriate patient positioning. Ultrasound guidance during an axillary incision at the projection of this lymph node allows direct access to the blue-stained sentinel lymph node. This approach reduces the extent of dissection and the need for channel tracking compared to the standard technique, resulting in a smaller incision, less tissue dissection, and shorter operative time.

This study evaluates whether ultrasound-guided projection of the first lymph node at the axillary entry during an axillary incision, followed by tracing the blue-stained lymphatic channel and identifying adjacent lymph nodes, reduces operative time and morbidity by minimizing dissection compared to the standard axillary hairline landmark approach.

ELIGIBILITY:
Inclusion Criteria:

* * Patients with clinical stage T1-T3 disease (tumor ≤5 cm), pN0-pN1 (one to three regional lymph nodes with micrometastases or metastases), and M0 (no distant metastasis) are eligible. Post-neoadjuvant yT1-T3, yN0-yN1, and M0 status are also eligible. All patients are undergoing axillary staging.
* Clinically negative axilla
* Written informed consent must be obtained prior to inclusio

Exclusion Criteria:

* Younger than 18 years
* Previous breast malignancy
* Pregnancy
* Pre-operative diagnosis of axillary lymph node metastases
* The presence of multiple clinically involved or suspicious lymph nodes
* Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for sentinel lymph node biopsy due to breast cancer at Antalya Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative assessment of surgical performance parameters. | Until completion of the sentinel lymph node procedure
  Measurements will include incision details and lymph node detection times.

CONTACTS AND LOCATIONS:
Overall Officials: Baris R KARAKAS, Assoc. Prof., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fenech M, Burke T, Arnett G, Tanner A, Werder N. Sonographic localisation of lymph nodes suspicious of metastatic breast cancer to surgical axillary levels. J Med Radiat Sci. 2025 Mar;72(1):119-138. doi: 10.1002/jmrs.840. Epub 2024 Nov 17. PMID 39552171
- [Background] Suami H, Pan WR, Mann GB, Taylor GI. The lymphatic anatomy of the breast and its implications for sentinel lymph node biopsy: a human cadaver study. Ann Surg Oncol. 2008 Mar;15(3):863-71. doi: 10.1245/s10434-007-9709-9. Epub 2007 Nov 28. PMID 18043970
- [Background] Gentilini OD, Botteri E, Sangalli C, Galimberti V, Porpiglia M, Agresti R, Luini A, Viale G, Cassano E, Peradze N, Toesca A, Massari G, Sacchini V, Munzone E, Leonardi MC, Cattadori F, Di Micco R, Esposito E, Sgarella A, Cattaneo S, Busani M, Dessena M, Bianchi A, Cretella E, Ripoll Orts F, Mueller M, Tinterri C, Chahuan Manzur BJ, Benedetto C, Veronesi P; SOUND Trial Group. Sentinel Lymph Node Biopsy vs No Axillary Surgery in Patients With Small Breast Cancer and Negative Results on Ultrasonography of Axillary Lymph Nodes: The SOUND Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1557-1564. doi: 10.1001/jamaoncol.2023.3759. PMID 37733364
- [Background] Veronesi U, Paganelli G, Galimberti V, Viale G, Zurrida S, Bedoni M, Costa A, de Cicco C, Geraghty JG, Luini A, Sacchini V, Veronesi P. Sentinel-node biopsy to avoid axillary dissection in breast cancer with clinically negative lymph-nodes. Lancet. 1997 Jun 28;349(9069):1864-7. doi: 10.1016/S0140-6736(97)01004-0. PMID 9217757
- [Background] Tanis PJ, Nieweg OE, Valdes Olmos RA, Kroon BB. Anatomy and physiology of lymphatic drainage of the breast from the perspective of sentinel node biopsy. J Am Coll Surg. 2001 Mar;192(3):399-409. doi: 10.1016/s1072-7515(00)00776-6. PMID 11245383